CLINICAL TRIAL: NCT07126743
Title: Accumulation Profiles of Specific Organic Pollutants in Adipose and Gastric Tissues of Bariatric Surgery Patients and Their Clinical Correlations With Obesity Severity
Brief Title: Organic Pollutant Build-Up in Body Fat and Stomach Tissue Linked to Obesity Levels
Status: Active, not recruiting | Type: Observational
Sponsor: Dong Peng (Other)
Responsible Party: Sponsor-Investigator, Dong Peng, Principal Investigator, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 2025-527-01
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Obesity &Amp; Overweight
Keywords: Metabolic syndrome; Organic pollutants; Obesity
MeSH Terms: conditions — Obesity; Overweight; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- obesity group: Adult patients diagnosed with obesity (body mass index ≥ 30 kg/m²) who are scheduled to undergo bariatric surgery for clinical indications, such as severe obesity or obesity-related comorbidities (e.g., type 2 diabetes, hypertension, dyslipidemia, or obstructive sleep apnea).
  The intervention of interest is the standardized collection of biological tissue samples during bariatric surgery. At the time of surgery, the investigators will obtain small samples of subcutaneous and visceral adipose tissue, as well as gastric tissue from the resected portion of the stomach, using sterile techniques. No additional incisions or surgical time beyond the standard bariatric procedure will be required.
  Interventions: Other: exposure to organic pollutant

INTERVENTIONS:
Other: exposure to organic pollutant — Small samples of subcutaneous and visceral adipose tissue will be analyzed for the presence and concentration of specific organic pollutants using validated analytical chemistry methods, such as gas chromatography-mass spectrometry (GC-MS) or liquid chromatography-mass spectrometry (LC-MS).

SUMMARY:
This study looks at whether certain environmental chemicals, called organic pollutants, build up in the body fat and stomach tissues of people with obesity who are having weight-loss (bariatric) surgery. These pollutants can come from things like plastics, pesticides, or industrial waste, and may affect health in different ways.

The investigators will measure the amount of these pollutants in tissue samples taken during surgery and see if the levels are different in people with mild, moderate, or severe obesity. By understanding these patterns, the investigators hope to learn more about how environmental factors may influence obesity and related health problems. The findings could help guide future prevention and treatment strategies for patients.

DETAILED DESCRIPTION:
Obesity is a complex health condition influenced by both lifestyle and environmental factors. Among these factors, persistent organic pollutants (POPs) - such as certain plastic-related chemicals, pesticides, and industrial byproducts - have raised growing concern due to their ability to accumulate in human tissues over time and potentially interfere with metabolism.

This study focuses on patients with obesity who are undergoing bariatric surgery. During surgery, the investigators will collect small samples of adipose (fat) tissue and gastric tissue under sterile conditions. These samples will be analyzed for the presence and concentration of specific organic pollutants using validated laboratory methods. The investigators will compare pollutant accumulation patterns across patients with varying levels of obesity severity, aiming to identify possible associations between pollutant burden and obesity-related clinical characteristics.

The results are expected to provide new insights into the environmental contributions to obesity, beyond diet and physical activity. By clarifying how pollutant accumulation in different tissues relates to obesity severity, the findings could help inform prevention strategies, refine clinical management, and highlight the need for targeted public health policies addressing environmental exposures.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years.
* BMI ≥30 kg/m² at screening (measured within 30 days before surgery).
* Scheduled for primary bariatric surgery (e.g., sleeve gastrectomy or Roux-en-Y gastric bypass) for clinical indications.
* Able to provide informed consent.
* Willing to allow intraoperative collection of subcutaneous/visceral adipose tissue and gastric tissue for pollutant analysis.
* Availability of basic preoperative clinical data (demographics, comorbidities, relevant labs).

Exclusion Criteria:

* Prior bariatric or major upper gastrointestinal surgery that alters stomach/anatomy relevant to sampling.
* Pregnant or breastfeeding at screening or on day of surgery.
* Active malignancy (excluding non-melanoma skin cancers) or ongoing systemic immunosuppressive therapy (e.g., chronic corticosteroids, biologics) within 3 months.
* Severe organ dysfunction: decompensated cirrhosis (Child-Pugh C) or eGFR <30 mL/min/1.73m².
* Acute infection or decompensated chronic illness that would preclude elective surgery per treating team.
* Documented high-level occupational or accidental chemical exposure within 6 months (e.g., pesticide poisoning) likely to bias tissue pollutant measurements.
* Participation in another interventional study expected to affect weight or metabolism within 3 months.
* Inadequate tissue obtainable at surgery for analysis (determined intraoperatively by the investigators).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients with obesity (BMI ≥30 kg/m²) scheduled to undergo primary bariatric surgery, including sleeve gastrectomy or Roux-en-Y gastric bypass, at participating surgical centers. Participants will represent a range of obesity severities (Class I-III) and may have obesity-related comorbidities such as type 2 diabetes, hypertension, dyslipidemia, or obstructive sleep apnea. All participants must be able to provide informed consent and agree to intraoperative collection of adipose and gastric tissue samples for organic pollutant analysis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Obesity Severity | At baseline (within 1 month before bariatric surgery).
  The investigators will assess obesity severity based on body mass index (BMI), calculated as body weight in kilograms divided by height in meters squared (kg/m²). BMI will be obtained using standardized measurements of height and weight during the preoperative evaluation. Obesity severity will be categorized according to World Health Organization (WHO) criteria (Class I: 30.0-34.9 kg/m², Class II: 35.0-39.9 kg/m², Class III: ≥ 40.0 kg/m²).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
individual participant data (IPD) will not be shared due to concerns regarding patient privacy, the sensitive nature of surgical and tissue analysis data, and applicable institutional and regulatory restrictions. Summary-level results will be made available in publications and presentations.